CLINICAL TRIAL: NCT02993289
Title: Is Detoxification Needed in Medication-overuse Headache?: A Randomized Controlled Trial of 3 Treatment Strategies
Brief Title: Is Detoxification Needed in Medication-overuse Headache?
Acronym: DEFINE3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Louise Carlsen, Medical doctor, PhD-student, Danish Headache Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-16029763
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Medication Overuse Headache
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Detoxification and pharmacological prophylactic treatment (Active Comparator): Group A: Two months detoxification program combined with pharmacological prophylactic treatment from start.
  Interventions: Other: Different well-known treatments
- Pharmacological prophylactic treatment (Active Comparator): Pharmacological prophylactic treatment from start without detoxification.
  Interventions: Other: Different well-known treatments
- Detoxification (Active Comparator): Two months detoxification program with postponed pharmacological prophylactic treatment after ended detoxification.
  Interventions: Other: Different well-known treatments
- Control group 1: Episodic migraine (No Intervention)
- Control group 2: Healthy volunteers (No Intervention)

INTERVENTIONS:
Other: Different well-known treatments
  Arms: Detoxification; Detoxification and pharmacological prophylactic treatment; Pharmacological prophylactic treatment

SUMMARY:
Medication-overuse headache (MOH) is a disabling condition, yet treatable. According to European guidelines and based on evidence, multidisciplinary detoxification is the first choice of treatment for MOH. However, consensus about the details in such detoxification programs is lacking. Contrary, other headache specialists believe more in treating chronic headache with medication overuse with single-therapy of prophylaxis and no withdrawal of acute medication, based on randomized controlled double-blinded placebo trial with prophylaxes. Only a single RCT has compared single-therapy with prophylaxis to detoxification. However there was no significant difference.

AIM:

1. To compare three different treatment protocols in order to improve the therapy of MOH.
2. To test several baseline variables for being potential predictors for good treatment outcome.
3. To examine the role of epigenetics in MOH.

ELIGIBILITY:
Patients with medication-overuse headache:

Inclusion Criteria:

* Confirmed MOH diagnosis according to the ICHD-III beta (1).
* Eligible for outpatient treatment based on type of medication overuse (without massive pure opioids and barbiturates overuse), and personal resources and motivation.
* Capable of completing headache diary/calendar.
* Age ≥ 18 years old and capable of providing informed consent.
* Medication-overuse headache based on initial tension-type headache (TTH) or migraine.
* Signed informed consent.

Exclusion Criteria:

* Severe physical illness or psychiatric disorders.
* Addiction to alcohol or other drugs.
* Current treatment with headache prophylaxis. Patients can be included minimum 5 weeks after stop of prophylaxis.
* Pregnancy, breastfeeding or planned pregnancy within the next 12 months.
* Inability to provide reliable information about medical history.

Criteria for Control group 1 - Episodic migraineurs:

* Episodic migraine, with/without concomitant tension-type headache, according to the ICHD-III beta.
* Headache days / month ≤ 6 at time of inclusion.
* Days with analgesics / month ≤ 6 at time of inclusion.
* Prophylactics are allowed.
* Age ≥ 18 years old.
* Ability to fill out headache calendar.
* No previous medication overuse.
* No significant co-morbid pain, physical or psychiatric disorders.
* No addiction to alcohol or drug-abuse.
* No pregnancy, breastfeeding or planned pregnancy within the next 12 months.

Criteria for Control group 2 - Healthy volunteers:

•≥ 2 days with headache in the past month at time of inclusion.

* Days with analgesics / month ≤ 6 at time of inclusion.
* Age ≥ 18 years old.
* No significant co-morbid pain, physical or psychiatric disorders.
* No addiction to alcohol or drug-abuse.
* No pregnancy, breastfeeding or planned pregnancy within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in headache days per month in group A and C compared to group B. | Six months follow-up

SECONDARY OUTCOMES:
Reduction in headache days per month | Two and 12 months follow-up and 4 years
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Reduction in days/month with use of analgesics and/or migraine medication. | Two, 6 and 12 months follow-up and 4 years
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Responders based on reduction in headache days / month (percentage with more than 30%, 50% and 75%). | Two, 6 and 12 months follow-up and 4 years
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Reduction in headache intensity. | Two, 6 and 12 months follow-up and 4 years
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  This outcome will be presented as 1) Total headache intensity per month, and as 2) Visual Analogue Scale (VAS).
Descriptive report of self-reported adverse effects of treatments. | Two, 6 and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Changes in Headache Under-Response to Treatment (HURT)-score. | Two, 6 and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Drop-out rate. | One, 2, 4, 6, 9 and 12 months follow-up and 4 years
Changes in Hospital Anxiety and Depression Scale (HADS). | Six and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Changes in Quality of Life (QoL) score. | Six and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Changes in Severity of Dependence Score (SDS). | Six and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Changes in Perceived Stress Score (PSS). | Twelve months follow-up.
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).
Patient's satisfaction questionnaire | Two, 6 and 12 months follow-up
  1. Group A and C versus group B.
  2. Group A (detoxification with prophylaxis) versus group C (detoxification with postponed prophylaxis).
  3. Group B (single-therapy with prophylaxis) versus group C (detoxification with postponed prophylaxis).

OTHER OUTCOMES:
Difference in DNA-profile between patients with MOH and controlgroups. | Baseline
Difference in methylation levels and RNA sequence analysis in patients with MOH undergoing treatment compared to controls. | From baseline to 6 months follow-up
Analysis of association between methylation levels and treatment outcome defined as 1) reduction in headache days per month at 6 months and 12 months and 2) percent of cured vs. percent of relapsers after 12 months. | At 6 and 12 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Carlsen LN, Hansen CS, Kogelman LJA, Werge TM, Ullum H, Bybjerg-Grauholm J, Hansen TF, Jensen RH. DNA-methylation and immunological response in medication overuse headache. Cephalalgia. 2023 Mar;43(3):3331024221147482. doi: 10.1177/03331024221147482. PMID 36786322
- [Derived] Carlsen LN, Munksgaard SB, Nielsen M, Engelstoft IMS, Westergaard ML, Bendtsen L, Jensen RH. Comparison of 3 Treatment Strategies for Medication Overuse Headache: A Randomized Clinical Trial. JAMA Neurol. 2020 Sep 1;77(9):1069-1078. doi: 10.1001/jamaneurol.2020.1179. PMID 32453406